CLINICAL TRIAL: NCT00917943
Title: Smoking Resumption-Prevention is Postpartum Women
Brief Title: Preventing Postpartum Return to Smoking
Acronym: Quit for Two
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00004337; 1R01NR009429-01A2 (NIH)
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Smoking
Keywords: smoking; pregnancy; counseling; prevention; tailored intervention; postpartum; women; cessation
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Counseling Intervention Arm (Experimental): Bio-behavioral and pregnancy-specific factors are used to triage women in the treatment arm to one of four levels of stepped-care that includes one in-person counseling session and at least one telephone session during pregnancy and from 6 to 11 telephone sessions over the first 9-months postpartum.
  Interventions: Behavioral: Tailored Counseling Intervention Arm
- Control Arm (No Intervention): Women randomized to the control arm receive the booklet, Forever Free for Baby and Me: A Guide to Remaining Smoke Free and usual prenatal and postpartum care.

INTERVENTIONS:
Behavioral: Tailored Counseling Intervention Arm — Study staff contact women when they are between 28 and 34 weeks pregnant, confirm their non-smoking status, and make an appointment to explain the study further, obtain written informed consent, conduct the risk assessment, and collect baseline data. Bio-behavioral and pregnancy-specific factors are used to triage women in the treatment arm to one of four levels of stepped-care that includes one in-person counseling session and at least one telephone session during pregnancy and from 6 to 11 telephone sessions over the first 9-months postpartum.
  Other Names: Nurse Counseling
  Arms: Tailored Counseling Intervention Arm

SUMMARY:
STUDY PURPOSE:

Aim 1. To assess the efficacy of an intervention in preventing or delaying postpartum smoking resumption among women who stop smoking during pregnancy.

Aim 2. To determine the association of baseline risk assessment variables (dependence, motivation, self-efficacy, concerns for the fetus, changes in sensory response to tobacco, depression, weight concerns, and partner/household smoking and support) with time to resumption.

A two-arm randomized controlled trial will be conducted. Women's risk for resumption will be assessed at 4 time-points.

1. Between 28 and 34 weeks of pregnancy
2. 6-weeks postpartum
3. 6-months postpartum
4. 12-months postpartum

Women who report not smoking at any of the assessment points will be asked to provide a saliva sample for analysis of tobacco constituents and a breath sample to assess carbon monoxide. Bio-behavioral and pregnancy-specific factors will be used to triage women to one of four levels of stepped-care that includes:

1. One in-person counseling session and at least one telephone session during pregnancy and from 6 to 11 telephone sessions over the first 9-months postpartum.
2. Risk profiles will be used to match the intervention to each woman's needs.
3. Women randomized to the control arm will receive the booklet, Forever Free for Baby and Me and usual prenatal and postpartum care.

We are recruiting 400 women for this study from 11 sites in the Durham/ Raleigh/ Chapel Hill NC area and Fayetteville NC.

DETAILED DESCRIPTION:
STUDY DESIGN:

A two-arm randomized controlled trial will be conducted. Women's risk for resumption will be assessed at 4 time-points.

1. Between 28 and 34 weeks of pregnancy
2. 6-weeks postpartum
3. 6-months postpartum
4. 12-months postpartum

Women who report not smoking at any of the assessment points will be asked to provide a saliva sample for analysis of tobacco constituents and a breath sample to assess carbon monoxide. Bio-behavioral and pregnancy-specific factors will be used to triage women to one of four levels of stepped-care that includes:

1. One in-person counseling session and at least one telephone session during pregnancy and from 6 to 11 telephone sessions over the first 9-months postpartum.
2. Risk profiles will be used to match the intervention to each woman's needs.
3. Women randomized to the control arm will receive the booklet, Forever Free for Baby and Me and usual prenatal and postpartum care.

SETTING:

We will recruit women for this study from 11 sites: Duke University Health Systems, Durham County Health Services, Person County Health Department, Orange County Health Department, Alamance County Health Department, Guilford County Health Department, Wake County Human Services, Durham OB, Harris and Smith (Durham), Womack Army Medical Center (WAMC), and Cape Fear Valley on the Fort Bragg Army Installation in Fayetteville, North Carolina.

SAMPLE:

The sample will be 400 women. To be eligible for the study women must be: 1) 18 years of age or older 2) speak English 3) registered for prenatal care and 4) have a history of smoking, defined as having smoked at least 100 cigarettes in their lifetimes and at least 5 cigarettes a day prior to becoming pregnant.

Eligible women will need to have been continuously abstinent from tobacco for at least 1 month prior to their risk assessment, which will occur between 28 and 34 weeks of pregnancy.

RECRUITMENT:

Initial Screening and Recruitment. At Duke and the Durham County Health Department, each week, all new obstetric patient charts are reviewed, and women with a history of tobacco use are sent a letter from their providers informing them of the study and asking them to call a toll-free number if they prefer not to be contacted about study participation. Women who do not call are contacted and screened for eligibility. At all other sites, nurses screen women and ask women to complete a contact sheet so that study staff can contact them.

Nurse Case Managers (NCM) contact women when they are between 28 and 34 weeks pregnant, confirm their non-smoking status, and make an appointment to explain the study further. Data Technicians obtain written consent, conduct risk assessment, and collect baseline data. Data is collected at the woman's prenatal clinic or at her home if she prefers or if her next prenatal appointment is outside our recruitment time frame.

Randomization procedures. Randomization occurs at each study site (Duke and WAMC). At each site, women are randomized to treatment or control condition with proportional risk categories represented in treatment and control groups. Women assigned to the control arm receive a tobacco control and family-centered relapse prevention booklet, Forever Free for Baby and Me.

RISK ASSESSMENT:

A risk profile is created for women based on the assessment of bio-behavioral (BB), pregnancy-specific (PS), and co-condition (CC) risk factors.

All follow-up data collection is conducted face-to-face by a blinded staff member (not Nurse Case Manager).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speak English
* Registered for prenatal care
* Have a history of smoking (defined as having smoked at least 100 cigarettes in their lifetimes and at least 5 cigarettes a day prior to becoming pregnant)
* Will need to have been continuously abstinent from tobacco for at least 1 month prior to their risk assessment
* Women will be eligible if they stopped smoking upon learning of their pregnancies and have been continuously abstinent (self-initiated quitters), or if they continued to smoke during the first few months of pregnancy but have been continuously abstinent from 24 to 28 weeks.

Exclusion Criteria:

* Any women who stopped smoking and resumed by the 34-week risk assessment will be ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of an intervention in preventing or delaying postpartum smoking resumption among women who stop smoking during pregnancy. | 12 months postpartum

SECONDARY OUTCOMES:
To determine the association of baseline risk assessment variables with time to resumption. | 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn I Pollak, PhD, Principal Investigator — Duke University; Evan Myers, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States